CLINICAL TRIAL: NCT04083196
Title: A Randomized, Blinded, Placebo-controlled Phase I Clinical Trial Evaluating the Safety and Preliminary Immunogenicity of a 11-valent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) in Chinese Women Aged 9-45 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry); Simoon Record Pharma Information Consulting Co., Ltd. (Industry); Guangxi Center for Disease Control and Prevention (Other Government); Beijing Kantorico Statistical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GXIRB2019-0030-1
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: HPV Infection; HPV-Related Cervical Carcinoma
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experiment group (Experimental): According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the experiment vaccine
  Interventions: Biological: 11-valent recombinant human papilloma virus vaccine (Hansenula polymorpha)
- placebo group (Placebo Comparator): According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 11-valent recombinant human papilloma virus vaccine (Hansenula polymorpha) — Injection vaccine produced by ChinaVaccineSerum ,containing HPV antigen protein, 270μg/1ml/bottle
  Arms: experiment group
Biological: Placebo — Placebo
  Arms: placebo group

SUMMARY:
A total of 90 Chinese women aged 9-45 years old were divided into three age groups: 27-45 years old, 18-26 years old, and 9-17 years old. The experimental group and the placebo group were randomly assigned in a ratio of 2:1. Sixty patients had a placebo group of 30 patients. All subjects enrolled in the upper arm deltoid muscle were injected with 3 doses of test vaccine or placebo according to the 0, 2, and 6 months immunization program.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chinese women aged 9-45 who can provide legal identification; 2. The legal guardian of the subject and/or subject has the ability to understand the research procedure and sign an informed consent form (a 9-17 year old subject signs an informed notification); 3).The legal guardian of the subject and / or subject has the ability to read, understand, fill in the journal card / contact card, and promise to participate in regular follow-up as required by the study; 4. Female children of childbearing age were not pregnant at the time of enrollment (negative urine pregnancy test), did not have lactation period and had no birth plan within the first 7 months after enrollment; effective contraceptive measures were taken within 2 weeks before enrollment in the study. And agree to continue to take effective contraceptive measures within the first 7 months after the study (effective contraceptives include: oral contraceptives, injection or embedding contraceptives, sustained release topical contraceptives, hormone patches, intrauterine devices) (IUD), sterilization, abstinence, condoms (male), diaphragms, cervical caps, etc.

Exclusion Criteria:

* 1. Previously vaccinated with commercially available HPV vaccines or planned to vaccinate commercially available HPV vaccines during the study period or have participated in HPV vaccine clinical trials and have received vaccine/placebo vaccination; 2. History of cervical lesions (such as cervical cancer screening abnormalities, history of CIN disease) or history of hysterectomy (vaginal or total abdominal hysterectomy) or history of pelvic radiation therapy; history of external genital diseases (such as vulvar epithelialization) Tumor, vaginal intraepithelial neoplasia and genital warts, etc. or acute genital infections (eg acute vaginitis, acute endometritis, acute salpingitis and oophoritis); or previous history of sexually transmitted diseases (including syphilis) Gonorrhea, genital warts, genital chlamydia infection, genital herpes, soft chancre, sexually transmitted lymphogranuloma, inguinal granuloma, etc.); 3. Have a history of severe allergies to any of the components of the test vaccine, including yeast, L-histidine, sodium chloride, aluminum hydroxide and water for injection, eg anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenia Sexual purpura, local allergic necrosis (Arthus reaction); or any previous history of serious side effects of vaccines or drugs, such as: allergies, urticaria, skin eczema, dyspnea, angioedema, etc.; 4. There is thrombocytopenia or other coagulopathy that can be a contraindication to intramuscular injection; 5. impaired immune function or has been diagnosed as having congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile Rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases; 6. no spleen or functional spleen, and no spleen or splenectomy caused by any condition; 7. has been diagnosed as having an infectious disease, such as: tuberculosis, hepatitis B, hepatitis C, etc.; 8. Before the enrollment, the physical examination was hypertension (systolic blood pressure ≥140mmHg and / or diastolic blood pressure ≥90mmHg) (applicable to 18-45 year olds); 9. suffering from severe cardiovascular disease (pulmonary heart disease, pulmonary edema), severe liver and kidney disease, and complications of diabetes; 10. 3 days before vaccination, suffering from acute illness or acute exacerbation of chronic disease; 11. have convulsions, epilepsy, encephalopathy, mental illness or family history; 12. Inactivated vaccine or recombinant vaccine within 14 days before vaccination, or vaccinated with any live vaccine within 28 days; 13. Participated in other gynecological related clinical trials within 6 months, participated in other research or unregistered products (drugs or vaccines) within 3 months, or planned to participate in other clinical studies after the clinical study was enrolled; 14. receive any immunoglobulin or blood product within 6 months prior to the first injection, or plan to receive such product by the 7th month of the study; 15. In the past 6 months, there have been immunosuppressive drugs, systemic medication for corticosteroids (≥2mg/kg/day, continuous use ≥14 days), but local medication (such as ointment, eye drops, inhalants) Or nasal spray), the topical medication should not exceed the recommended dose in the instructions or have any systemic exposure signs; 16. The body temperature before inoculation on the day of enrollment> 37.0 ° C (armpit temperature); 17. Before the first dose is vaccinated, the laboratory test indicators specified in the program are abnormal and clinically determined by the clinician; 18. plan to move out of the country before the end of the study or leave the local area for a long time during the scheduled study visit; 19. The investigator believes that the subject has any condition that may interfere with the assessment of the purpose of the study.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
AE of local and systemic reactions within 30 minutes after each dose | 30 min
All active AEs within 0-7 days after each dose | 7 days
  Active AE: Local and systemic adverse reactions occurring within 0-7 days after each dose of vaccination
All non-active collection AEs within 0-30 days after each dose | 30 days
  Adverse events other than active AE include solicitation adverse events reported in addition to the specified solicitation time window
All SAEs within 6 months after the first dose is vaccinated | 6 months

SECONDARY OUTCOMES:
Geometric mean titer of neutralizing antibodies against HPV types 6, 11, 16, 18, 31, 33, 45, 52, 58, 59 and 68 30 days after full immunization (Geometric Mean Titer, GMT) | 7 months
Neutralizing antibody positive rate of anti-HPV6, 11, 16, 18, 31, 33, 45, 52, 58, 59 and 68 antibodies 30 days after full immunization | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Liuzhou Center for Disease Control and Prevention, Liuchow, Guangxi, China

IPD SHARING:
Plan to Share IPD: No